CLINICAL TRIAL: NCT04932395
Title: An Adaptive Enrichment Designed, Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Trial of Anshen Buxin Liuwei Pills in the Treatment of Cardiac Neurosis
Brief Title: Anshen Buxin Liuwei Pills for the Treatment of Cardiac Neurosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government); Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASBXLWW V2.0
Record Dates: First submitted 2021-06-12; First posted 2021-06-21 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Cardiac Neurosis
MeSH Terms: conditions — Neurocirculatory Asthenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anshen Buxin Liuwei Pills (Experimental): 15 pills/time, 2 times/day, orally，for 8 weeks
  Interventions: Drug: Anshen Buxin Liuwei Pill
- Placebo (Placebo Comparator): 15 pills/time, 2 times/day, orally. for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anshen Buxin Liuwei Pill — 15 capsules/time, 2 times/day, orally.
  Arms: Anshen Buxin Liuwei Pills
Drug: Placebo — Placebo simulated as the Anshen Buxin Liuwei Pills with same appearance，smell and taste,15 capsules/time, 2 times/day, orally.
  Arms: Placebo

SUMMARY:
This study aims to assess the effect and safety of the traditional Mongolian medicine Anshen Buxin Liuwei Pill for the treatment of cardiac neurosis.

DETAILED DESCRIPTION:
Cardiac neurosis is a group of symptoms characterized by the coexistence of cardiovascular disease related symptoms and nervous system disorders. Anshen Buxin Liuwei Pill is a kind of traditional Mongolian medicine for the treatment of cardiac neurosis. This study aims to evaluate the effect and safety of Anshen Buxin Liuwei Pill for cardiac neurosis in a prospective, randomized, double-blind, placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, ≤75 years old;
* Meet the diagnostic criteria for cardiac neurosis: the patient has palpitations, precordial pain, chest tightness, shortness of breath, dyspnea, dizziness, insomnia and dreaminess, cold hands and feet, hyperhidrosis and other cardiovascular symptoms and neurological disorders;
* Meet the diagnostic criteria of Heyisheng type palpitations in Mongolian medicine;
* There is no objective diagnosis of coronary heart disease (in accordance with any of the following): ①The activity flat test is negative; ② Coronary angiography or coronary CTA suggests that the lumen stenosis is ≤50%; ③ Exercise or drug load radionuclide examination results suggest no myocardial ischemia;
* The patient did not take anti-anxiety and depression drugs or psychotropic drugs within 2 weeks before enrollment;
* agrees to voluntarily participate in the study and signs an informed consent form .

Exclusion Criteria:

* Accompanied by organic heart disease, severe cardiopulmonary insufficiency;
* Poor hypertension control (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg after treatment);
* Those with malignant arrhythmia;
* Those who use pacemakers;
* Patients with hyperthyroidism;
* Combined with severe liver and kidney damage (ALT, AST or TBIL> 2 times the upper limit of the normal reference value, or Cr> 1.5 times the upper limit of the normal reference value);
* People with serious primary diseases such as hematopoietic system or mental illness;
* SAS≥70;
* SDS≥73;
* Accompanying any other serious diseases or conditions such as malignant tumors;
* Women during pregnancy and lactation;
* People with allergies or allergies to the known ingredients of the research drug;
* Participated in other clinical research in the past 3 months;
* According to the judgment of the investigator, the subject is not suitable for research observation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Palpitation with Heyisheng Type Symptoms Scale in Mongolian Medicine | 8 weeks
  The scale is to record the symptoms of palpitation with Heyisheng Type in Mongolian Medicine, which is also usually seen in cardiac neurosis. This scale includes two domain: the primary symptoms and the secondary symptoms. The domain of the primary symptoms includes palpitations, chest tightness, chest pain, insomnia, and restlessness using the evaluating 4-Grade scales (Normal:0; Mild:3; Moderate:6 and Severe:9), while the domain of the secondary symptoms includes dizziness, like to sigh, easy to startle, tinnitus, blurred vision, fatigue, sweating, irritability, using the evaluating 4-Grade scales (Normal:0; Mild:1; Moderate:2 and Severe:3).

SECONDARY OUTCOMES:
Cardiac autonomic nervous function | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks.
  The cardiac autonomic nervous function was evaluated by detecting the difference in heart rate per minute between standing and lying positions using RR interval in lead Ⅱ ECG.
Cardiac Neurosis Symptom Self-rating Scale | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks.
  This self-rating scale was used to evaluate the main symptoms in cardiac neurosis, including palpitations, chest tightness, chest pain, hyperhidrosis, insomnia, irritability, with each symptom evaluated via a 4-grading scale (normal:0 points, mild: 1 point, moderate: 2 points, severe:3 points
Self-rating depression scale (SDS) | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks.
  The Self-Rating Depression Scale (SDS) which was designed by Zung was adopted to assess participants' symptoms of depression during the past week. The SDS assesses depressive symptoms on a four-point scale ranging from "a little of the time" (value = 1) to "most of the time" (value = 4). The standard score is equal to the integer portion of 1.25 times the total score. The standard score of SDS is interpreted as: normal (≤52), mild (53-62), moderate (63-72), and severe (≥73).
Self-rating Anxiety Scale (SAS) | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks.
  The SAS is a 20-item measure developed to assess the frequency of anxiety symptoms based on diagnostic conceptualizations. It consists primarily of somatic symptoms. The respondent indicates how often he or she has experienced each symptom on a 4-point Likert scale consisting of "one or a little of the time" (coded as 1), "some of the time" (coded as 2), "good part of the time" (coded as 3), and "most or all of the time" (coded as 4). Items 5, 9, 13, 16, and 19 are reversed scored and total scores on the SAS range from 0 to 80.
Pittsburgh Sleep Scale Score | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks.
  The PSQI comprises 19 self-evaluation items, among which 18 items generate 7 components. Each component is graded from 0 to 3, and the cumulative score of each component is the total score of PSQI, which ranges from 0 to 21.
Consumption of estazolam | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks.
  If the patient has a moderate or above anxiety and depression state and is intolerable, he could be given a short-term sedative and hypnotic drug,estazolam, and the frequency and dose of estazolam should be recorded in the patient's diary
hypersensitive C-reactive protein (hs-CRP) | Baseline, 4 weeks, 8 weeks
  hs-CRP is used to evaluate the level of systemic inflammation in the patients with cardiac neurosis.
The level of serotonin | Baseline, 4 weeks, 8 weeks
  The decrease of serotonin is reported in the patients with cardiac neurosis. The level of serotonin could be used to evaluate the effect for cardiac neurosis.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Nanyang First People's Hospital, Nanyang, Henan
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - The First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - Inner Mongolia International Mongolian Hospital, Hohhot, Inner Mongolia
  - Kunshan First People's Hospital, Kunshan, Jiangsu
  - The Second Affiliated Hospital of Shandong University of Chinese Medicine, Jinan, Shandong